CLINICAL TRIAL: NCT01149902
Title: Phase I Study of Chemo-Immunotherapy in Patients With Relapsed and Refractory Head and Neck Squamous Cell Carcinoma
Brief Title: Study of Chemo-Immunotherapy in Head and Neck Cancer Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Yamanashi (Other)
Responsible Party: Keisuke Masuyama, Professor, Department of Otolaryngology-Head and Neck Surgery, University of Yamanashi, Faculty of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 631
Record Dates: First submitted 2010-06-22; First posted 2010-06-24 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2010-06

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cyclophosphamide; Docetaxel; Picibanil

INTERVENTIONS:
Biological: Cyclophosphamide, Docetaxel, Dendritic cells, OK-432 — Cyclophosphamide 50mg/day, day1-7 and 22-28 Docetaxel 30mg/m2, day6 and 27 OK-432 5KE/day, day7,14,28,35

SUMMARY:
The purpose of this study is to determine safety and feasibility of Chemo-Immunotherapy using cyclophosphamide, docetaxel, OK-432, and autologous immature dendritic cells for patients with relapsed and refractory head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with relapsed and refractory head and neck squamous cell carcinoma
2. 20 years and older
3. ECOG performance status 0-1
4. More than 4 weeks must have elapsed from the time of radiation therapy and the last dose of chemotherapy
5. Tumor lesions are accessible to intratumoral dendritic cells injection
6. Patients who are able to do oral ingestion
7. Patients must have normal organ and marrow functions as follows:

   * Hb>9.0 mg/dl
   * Ht>25%
   * WBC>4000/mm3
   * Platelet count>100,000/mm3
   * T-Bil<1.5mg/dl
   * GOT<x2.5 institutional upper limit of normal
   * GPT<x2.5 institutional upper limit of normal
   * Creatinin<1.5mg/dl
8. signed informed consent

Exclusion Criteria:

1. Less than 20 years
2. Patients who test positive for Hepatitis B virus, Hepatitis C virus or HIV.
3. Patients with clinically active infection
4. Patients with uncontrolled concurrent illness including cardiovascular disease, pulmonary disease, and bleeding tendency
5. Concomitant malignant diseases, brain metastases
6. Psychiatric illness
7. Treatment with steroids
8. Decision of unsuitableness by physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
The safety and feasibility of chemo-immunotherapy | 1 year

SECONDARY OUTCOMES:
The number and function of immune effector cells in treated patients | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Umiversity of Yamanashi Hospital, Chūō, Yamanashi, Japan